CLINICAL TRIAL: NCT05486273
Title: Evaluation of the Impact of Sports-inspired Onco-coaching on Health-related Quality's Life of the Patients in Cancer Remission After Allogeneic Transplantation of Hematopoietic Stem Cells : a Randomized Controlled Trial REBOND2-IPC 2022-009
Brief Title: Evaluation of the Impact of Sports-inspired Onco-coaching on Health-related Quality's Life of the Patients in Cancer Remission After Allogeneic Transplantation of Hematopoietic Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REBOND2-IPC 2022-009
Record Dates: First submitted 2022-07-28; First posted 2022-08-03 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-08

CONDITIONS: Hematological Cancer
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: They will be randomized unequally (2:1) into one of the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Groupe OC (Onco-Coaching) (Experimental): You will be offered 6 coaching sessions at a rate of one session per month. The first session will take place in the month following your inclusion in the study.
  The study also includes the evaluation, by quality of life questionnaires, of the well-being variables (Self-efficacy, Capabilities, PANAS and Life Satisfaction, Hope, Anxiety and Depression in hospital, Subjective well-being and Health benefit).
  They should be completed at the time of inclusion in the protocol at 1, 3, 6, 9 and 12 months after inclusion. The purpose of these interviews is to ask more specific questions about the impact of the program.
  Interventions: Other: interviews with coachs, semi-structured interviews and questionnaires
- Groupe C (Contrôle) (Active Comparator): the patient will have standard management including also questionnaires and semi-structured interviews within the same time frame as the experimental arm.
  Interventions: Other: semi-structured interviews and questionnaires

INTERVENTIONS:
Other: interviews with coachs, semi-structured interviews and questionnaires — You will be offered 6 coaching sessions at a rate of one session per month and the first interview will be conducted on the day of inclusion or within one month of inclusion, the others will take place at R6 and R12. Questionnaires will be administered on the day of inclusion and then at R1, R6, R9 and R12. RO is the day of inclusion and it corresponds to M3 (3 months post transplant)
  Arms: Groupe OC (Onco-Coaching)
Other: semi-structured interviews and questionnaires — The first interview will be conducted on the day of inclusion or within one month of inclusion, the others will take place at R6 and R12.Questionnaires will be administered on the day of inclusion and then at R1, R6, R9 and R12. RO is the day of inclusion and it corresponds to M3 (3 months post transplant)
  Arms: Groupe C (Contrôle)

SUMMARY:
To measure the impact of a coaching program on the patient's health-related quality of life 15 months post-transplant (M15/R12).

DETAILED DESCRIPTION:
After signing the consent form and validating the inclusion and non-inclusion criteria, patients will be included in the study. They will be randomized unequally (2:1) into one of the study groups:

* OC (Onco-Coaching) group: patients will undergo onco-coaching sessions at a rate of 1 session/month until 6 months post-inclusion (M9/R6). 73 patients will be randomized in this group
* Group C (Control): Patients will not receive onco-coaching follow-up, but will be able to benefit from classical management in full autonomy. 35 patients will be randomized in this group

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age and have a good understanding and practice of the French language,
2. Have been treated by an allogeneic hematopoietic stem cell transplant
3. Signed consent to participate,
4. Affiliation with a social security plan, or beneficiary of such a plan.

Exclusion Criteria:

1. Patients under treatment for complications (infections, GvHD,...) except patients with cGvHD requiring corticosteroid therapy less than or equal to 1 mg/kg daily
2. Patient with progressive or relapsing hematological disease,
3. Person in an emergency situation, adult under legal protection (guardianship, curatorship or safeguard of justice), or unable to express his/her consent,
4. Person requiring psychotherapeutic care
5. Impossibility to submit to the follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
To measure the impact of a coaching program on the patient's health-related quality of life 15 months post-transplant (M15/R12). | from inclusion(RO=M3) to R12( Month 15 =12 month post inclusion)
  evolution over time of the FACT-BMT( Functional Assessment of Cancer Therapy - Bone Marrow Transplantation) score during the first 15 months after transplantation the highest score corresponds to a worse condition of the patient.the value are between 0 and 200

SECONDARY OUTCOMES:
To measure the impact of a coaching program on patient quality of life sub-dimensions 15 months post-transplant (M15/R12). | from inclusion(RO=M3) to R12(Month15 =12 month post inclusion)
  evolution of the FACT-BMT(Functional Assessment of Cancer Therapy - Bone Marrow Transplantation) score up to R12 evolution over time of sub-scores related to physical well-being, social well-being, functional well-being and relationship with the physician.the quality of life is a questionnaire with scores ranging from 5 to 20
Measure the impact of a coaching program on the patient's empowerment (capabilities, subjective well-being, hope and self-efficacy). | from inclusion(RO=M3) to R12(Month15 =12 month post inclusion)
  evolution over time of self-efficacy (the higher the score, the better the efficiency), capability, subjective well-being and hope scores
Measure the impact of a coaching program on reducing emotional distress. | from inclusion(RO=M3) to R12(Month 15 =12 month post inclusion)
  changes over time in HADS scores (Hospital Anxiety and Depression Scale)the highest score corresponds to high anxiety and depression the value are between 0 and 21 but if the patient has a score higher than 11, he is suffering from anxiety or depression
Evaluate the cost-utility of the coaching program. | from inclusion(RO=M3) to R12(Month15 =12 month post inclusion)
  incremental cost-effectiveness ratio (QALYs)
Assess correlations between quality of life and patient empowerment | from inclusion(RO=M3) to R12(Month15 =12 month post inclusion)
  evolution over time of the patient's speech (semi-directive interviews)
Assess the overall survival of participants | from inclusion(RO=M3) to R12(Month15 =12 month post inclusion)
  measure the overall survival rate at M15/R12

CONTACTS AND LOCATIONS:
Overall Officials: Didier BLAISE, Pr, Principal Investigator — Institut Paoli-Calmettes

IPD SHARING:
Plan to Share IPD: No